CLINICAL TRIAL: NCT03462940
Title: Pilot Study of The Effects of Tauroursodeoxycholic Acid (TUDCA) on Endothelial Function in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of TUDCA on Endothelial Function in Type 2 DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted due to low enrollment exacerbated by COVID-19.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-35009
Record Dates: First submitted 2018-02-27; First posted 2018-03-13 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Response; Endothelial Dysfunction
Keywords: Tauroursodeoxycholic acid (TUDCA); Endothelial function in humans; Endoplasmic Reticulum Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ursodoxicoltaurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TUDCA Group (Experimental): All subjects will receive 500 mg/day in a one week run-in period and then 1750 mg/day in one week treatment period of of the nutritional supplement Tauroursodeoxycholic acid (TUDCA).
  Interventions: Dietary Supplement: Tauroursodeoxycholic acid

INTERVENTIONS:
Dietary Supplement: Tauroursodeoxycholic acid — Tauroursodeoxycholic acid is an ambiphilic bile acid. It is the taurine conjugate form of ursodeoxycholic acid.
  Other Names: TUDCA

SUMMARY:
The pilot study is designed to investigate the acute and chronic effects of the diet supplement tauroursodeoxycholic acid (TUDCA) on endothelial function in participants with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a pilot study designed to investigate the effect of two doses of TUDCA on endothelial function.All subjects will receive 500 mg/day in a one week run-in period and then 1750 mg/day in one week treatment period. The study will consist of four visits (screening visit and three study visits), and last up to 2 weeks for individual subjects, depending on the time between visits. It is estimated that the study will last two years from IRB approval through data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus defined as fasting glucose greater than or equal to 120 mg/dL, HgA1C ≥6.5% or ongoing treatment with hypoglycemic medication.
* Willing to give written informed consent and able to understand, to participate in and to comply with the study requirements.

Exclusion Criteria:

* Women lactating or pregnant. All women with childbearing potential will undergo a urine pregnancy test at each visit to exclude pregnancy.
* Treatment with an investigational product within the last 30 days.
* Clinically evident major illness of other organ systems, including end-stage cancer, renal failure, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
* Inability to provide informed consent.
* Clinical instability that would preclude withholding medications as determined by the study physician.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Change in vascular function | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  Endothelium -dependent flow-mediated dilation of the brachial artery by ultrasound and fingertip tonometry at baseline and 5-minute cuff occlusion of the upper arm.

SECONDARY OUTCOMES:
Change in endoplasmic reticulum stress | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  Endothelial cells will be collected utilizing a J-wire inserted into an arm vein with an 18 gauge catheter using sterile technique and local anesthesia. ER stress will be measured by the study of early and chronic markers of ER stress activation by western blotting and PCR techniques.
Change in endothelial function | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  Endothelial cells will be collected utilizing a J-wire inserted into an arm vein with an 18 gauge catheter using sterile technique and local anesthesia. Endothelial function will be measured by the study of endothelial nitric oxide synthase activation and nitric oxide production
Change in fasting glucose | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  The blood sample will be processed to measure fasting glucose levels
Change in insulin levels | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  The blood sample will be processed to measure insulin levels
Change in lipid levels | before and 4 hours after TUDCA treatment at the screening and 3 study visits during a 2 week period
  The blood sample will be processed to measure lipids levels including total cholesterol, LDL, HDL and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No